CLINICAL TRIAL: NCT04652050
Title: Evaluation of Tolsura When Used as Prophylaxis After Lung Transplantation
Acronym: Tolsura
Status: Withdrawn | Type: Observational
Why Stopped: Patients are not interested to participate
Sponsor: Hong Nguyen (Other)
Responsible Party: Sponsor-Investigator, Hong Nguyen, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY20080119
Record Dates: First submitted 2020-11-23; First posted 2020-12-03 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Lung Transplant Infection
Keywords: lung transplant
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — excess biological samples collected as part of the patient's clinical care will be obtained if available for further testing/analysis for amounts of Tolsura
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- lung transplants: Lung transplants on Tolsura for infection
  Interventions: Drug: Tolsura

INTERVENTIONS:
Drug: Tolsura — Patients fulfilling the inclusion criteria (see above) and placed on Tolsura for prophylaxis, and signed informed consent to participate in this study will be part of the study.

SUMMARY:
This is a single-center, observational study of Tolsura PK sampling in lung transplant recipients

DETAILED DESCRIPTION:
Patients who are receiving Tolsura as part of their clinical care will be asked to enroll and EMR data and excess biological samples will be collected

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* hospitalized at UPMC
* placed on Tolsura prophylactically by clinical team
* patients who have had or will have a lung transplant.

Exclusion Criteria:

* redo lung transplant
* recipient with dual liver-lung transplant
* patients with previous history of SOT
* including other organ transplantation
* patients with known pre-transplant colonization with moulds resistant to azoles
* patients with intra-transplant positive cultures for moulds in either transplant recipient or his/her donor
* patients with a history of hypersensitivity reaction to an azole agent
* patients who are kept NPO (nothing by mouth, including meds)
* recipients or donor with HepC PCR positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung transplants on Tolsura that meet entry criteria
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
PK Sampling-measure amount of drug in system | one day PK sampling
  blood samples around a dosing of Tolsura to determine maximum plasma concentration

SECONDARY OUTCOMES:
rates of infection post treatment with Tolsura | 6 months
  follow lung transplant recipients till end of Tolsura treatment and determine rates of infection for as well as type of infections

CONTACTS AND LOCATIONS:
Overall Officials: Hong Nguyen, MD, Principal Investigator — UPMC and PITT
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
If data is shared all data provided de identified using alpha/numeric codes and MTA and/or DUA's will be in put in place prior to sharing